CLINICAL TRIAL: NCT01667250
Title: Non-Invasive Neurostimulation of the Vagus Nerve With the GammaCore Device for the Prevention of Chronic Migraine
Brief Title: Non-Invasive Neurostimulation for the Prevention of Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M-US-02
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Chronic Migraine
Keywords: vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; chronic migraine; migraine; non invasive; gammacore
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GammaCore Active Device (Active Comparator): Subjects will use an Active GammaCore Device
  Interventions: Device: GammaCore Active Device
- GammaCore Sham Device (Sham Comparator): Subjects who treat with the gammacore sham device in Phase 2 will receive the active gammacore treatment during phase 3 (active treatment) of this study.
  Interventions: Device: GammaCore Active Device; Device: GammaCore Sham Device

INTERVENTIONS:
Device: GammaCore Active Device
Device: GammaCore Sham Device
  Arms: GammaCore Sham Device

SUMMARY:
The purpose of this multi-center, prospective, double-blind, randomized, sham-controlled pilot study is to study feasibility and collect preliminary clinical data related to the safety and clinical benefits of daily use of non-invasive vagal nerve stimulation with the GammaCore device for the prevention of chronic migraine, and to support the development and approval of a larger pivotal study.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 18 and 65 years.
* Has been previously diagnosed as suffering from migraine, in accordance with the ICHD-2 Classification criteria (2nd), with or without aura.
* Experiences at least 15 headache days per month (over the last 3 months).
* Has age of onset of migraine less than 50 years old.
* Agrees not to use any migraine prevention treatments (including Botox injections) and/or medications (exclusive of medications taken for acute relief of migraine symptoms).
* Is able to provide written Informed Consent
* Agrees to refrain from changing the type or dosage of any prophylactic medications for indications other than chronic migraine that in the opinion of the clinician may interfere with the study

Exclusion Criteria:

* Has a history of aneurysm, intracranial hemorrhage, brain tumors or significant head trauma.
* Has a lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the GammaCore treatment site.
* Has known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of TIA or CVA), congestive heart failure (CHF), known severe coronary artery disease or recent myocardial infarction.
* Has an abnormal baseline ECG (e.g. second and third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction)
* Has had a previous bilateral, right, or left cervical vagotomy.
* Has uncontrolled high blood pressure.
* Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* Has a history of carotid endarterectomy or vascular neck surgery on the right side.
* Has been implanted with metal cervical spine hardware or has a metallic implant near the GammaCore stimulation site.
* Has a recent or repeated history of syncope.
* Has a recent or repeated history of seizure.
* Has a known history or suspicion of substance abuse or addiction.
* Has had a surgery for migraine prevention.
* Has received Botox injections for migraine prevention within the past 6 months.
* Has taken medications for migraine prophylaxis in the previous 30 days.
* In the opinion of the investigator/research staff the subject is incapable of operating the GammaCore device as intended and performing the data collection procedures.
* Is pregnant, nursing, thinking of becoming pregnant in the next 9 months, or of childbearing years and is unwilling to use an accepted form of birth control.
* Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).
* Is a relative of or an employee of the investigator or the clinical study site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSF Headache Center, San Francisco, California
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Headache Care Center, Springfield, Missouri
  - Montefiore Headache Center, The Bronx, New York
  - Carolina Headache Institute, Chapel Hill, North Carolina
  - Thomas Jefferson Headache Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Silberstein SD, Calhoun AH, Lipton RB, Grosberg BM, Cady RK, Dorlas S, Simmons KA, Mullin C, Liebler EJ, Goadsby PJ, Saper JR; EVENT Study Group. Chronic migraine headache prevention with noninvasive vagus nerve stimulation: The EVENT study. Neurology. 2016 Aug 2;87(5):529-38. doi: 10.1212/WNL.0000000000002918. Epub 2016 Jul 13. PMID 27412146
- See also: Effect of noninvasive vagus nerve stimulation on acute migraine: An open-label pilot study — https://www.ncbi.nlm.nih.gov/pubmed/24607501

RESULTS

PARTICIPANT FLOW:
Groups:
- GammaCore Active Device: Subjects will use an Active GammaCore Device
  GammaCore Active Device
- No Treatment (run-in, Enrollment Period): The run-in period was 1 month, Subject who did not fulfill the inclusion and/or exclusion criteria was not randomized to the treatment groups
Period: Run-in (no Treatment)
Arm/Group | GammaCore Active Device | GammaCore Sham Device | No Treatment (run-in, Enrollment Period)
Started | 0 | 0 | 73
Completed | 0 | 0 | 59
Not Completed | 0 | 0 | 14
Period: Randomised Period
Arm/Group | GammaCore Active Device | GammaCore Sham Device | No Treatment (run-in, Enrollment Period)
Started | 30 | 29 | 0
Completed | 29 | 28 | 0
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | GammaCore Active Device | GammaCore Sham Device | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Full Range); unit: years] | 39.7 [18.2 to 65.2] | 41.0 [20.0 to 60.9] | 40 [18.2 to 65.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 25 | 51
  Black | 3 | 0 | 3
  Hispanic | 1 | 2 | 3
  Other | 0 | 1 | 1
  Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants With Adverse Events
Description: Safety was assessed by collecting Adverse Effects
Time Frame: Up to 8 weeks - duration of the Randomized period
Population: Randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | GammaCore Active Device | GammaCore Sham Device
Number analyzed (Participants) | 30 | 29
Participants | 6 | 5

2. Secondary Outcome: Mean Change in Headache Days
Description: Mean change in headache days. Change between 4 week run in period to the 8 weeks randomized period.
Time Frame: Run-in period (4 weeks no treatment) and Randomized period (8 weeks)
Population: Data missing for 1 subject in each treatment group
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GammaCore Active Device | GammaCore Sham Device
Number analyzed (Participants) | 29 | 28
days | -1.5 (5.92) | -0.2 (3.52)

3. Secondary Outcome: Total Number of Headache Days Per Arm With Peak Severity of Mild, Moderate, or Severe
Description: Peak severity per headache day was reported each headache day in the subject diary. Pain was reported as mild, moderate or severe. Whereas as mild = least severe and severe = most severe.
Time Frame: Run-in (4 weeks no treatment) and Randomized (8 weeks)
Population: Randomized population
Measure: Number; unit: Headache days
Arm/Group | GammaCore Active Device | GammaCore Sham Device
Number analyzed (Participants) | 30 | 29
Headache days
  Run-in Mild | 167 | 131
  Run-in Moderate | 297 | 330
  Run-in Severe | 190 | 225
  Randomized Mild | 297 | 250
  Randomized Moderate | 443 | 511
  Randomized Severe | 274 | 395

4. Secondary Outcome: Use of Pain Relief Medication
Description: All abortive headache medication taken during randomized period
Time Frame: Randomized period - 8 weeks
Population: Randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | GammaCore Active Device | GammaCore Sham Device
Number analyzed (Participants) | 30 | 29
Participants
  Subjects taking abortive medication | 26 | 25
  Subjects taking no abortive medication | 3 | 3
  Subjects with no data | 1 | 1

5. Secondary Outcome: Mean Change in Quality of Life Short Form Survey (SF-12)
Description: The Quality of Life Short Form Survey (SF-12) is a multipurpose short form survey with 12 questions that are combined, scored and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. The SF-12 is weighted and summed to provide easily interpretable scales for physical and mental health. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of the twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
  SF-12 were recorded in the subject diary at the Phase 1 follow-up visit (week 4) and during Phase 2 randomized period at week 4 and week 8.
Time Frame: Run-in (4 weeks) and Randomized period (8 weeks)
Population: Randomized period
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GammaCore Active Device | GammaCore Sham Device
Number analyzed (Participants) | 30 | 29
Score on a scale
  Run-in PCS score | 40.9 (9.62) | 35.6 (10.46)
  Randomized period PCS score 4 weeks | 44.0 (9.25) | 37.5 (12.73)
  Randomized period PCS scores 8 weeks | 45.3 (8.01) | 38.0 (10.67)
  Run-in MCS scores | 44.5 (11.41) | 45.8 (10.55)
  Randomized period MCS scores 4 weeks | 44.7 (10.53) | 45.8 (11.71)
  Randomized period MCS scores 8 weeks | 46.5 (9.95) | 44.3 (12.24)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks - duration of the Randomized period
Arm/Group | GammaCore Active Device | GammaCore Sham Device
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/29
Other Adverse Events (participants affected / at risk) | 6/30 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GammaCore Active Device (N=30) | GammaCore Sham Device (N=29)
Worsening of Headache Pain (Nervous system disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GammaCore Active Device (N=30) | GammaCore Sham Device (N=29)
Altered sensations (brain zaps) (Nervous system disorders) | 1 (1) | 0 (0)
Migratory Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Right arm (hand) tremor (Nervous system disorders) | 1 (1) | 0 (0)
Right eye twitching (Nervous system disorders) | 2 (2) | 0 (0)
Lip twiching (Nervous system disorders) | 1 (1) | 0 (0)
Intermittent Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Exacerbated migraine (Nervous system disorders) | 1 (1) | 2 (2)
Lip numbness (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blister at treatment site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
General malaise (Infections and infestations) | 1 (1) | 0 (0)
Atypical migraine pain with associated blackouts (Nervous system disorders) | 0 (0) | 1 (1)
Sore throat (Infections and infestations) | 0 (0) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash at treatment site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mild pains in head and right arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Open label - phase 3
Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Open label - phase 3
Worsening of migraine (Nervous system disorders) | 1 (1) | 0 (0) — Open label - phase 3
Blisters at treatment site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Open label - phase 3
Rash/Blister at treatment site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Open label - phase 3
Redness at treatment site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Open label - phase 3
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Open label - phase 3
Severe migraine (Nervous system disorders) | 1 (1) | 0 (0) — Open label - phase 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less